CLINICAL TRIAL: NCT05960695
Title: The Effect of Relaxation and Stretching Exercises on Pain and Quality of Life in Women With Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pyeditepe
Record Dates: First submitted 2023-05-26; First posted 2023-07-27 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Pain; Exercise; Stretching
MeSH Terms: conditions — Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: The volunteers who met the inclusion criteria were divided into 2 groups. The patients have informed about 2 different groups, but they were not told which of them. Stretching exercises were taught regardless of which group the patients were in. In addition, relaxation exercises were taught to the patients in the stretching+relaxation group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Experimental Group (Experimental): The experimental group will be given both stretching and relaxation exercises. Among the stretching exercises, iliopsoas, adductor, and hamstring stretches will be taught.
  Deep breathing exercises will be taught as relaxation exercises. Participants will repeat the stretches 3 times a week with 3 repetitions of each stretch for 20 seconds.
  Interventions: Other: Stretching; Other: Relaxation
- The Control group (Active Comparator): The Control group will be given only stretching exercises. Among the stretching exercises, iliopsoas, adductor, and hamstring stretches will be taught.
  Participants will repeat the stretches 3 times a week with 3 repetitions of each stretch for 20 seconds.
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Stretching — Among the stretching exercises, iliopsoas, adductor, and hamstring stretches will be taught. Participants will repeat the stretches 3 times a week with 3 repetitions of each stretch for 20 seconds. The exercises will be done online by the physiotherapist.
  The experimental group will be given both stretching and relaxation exercises. The Control group will be given only stretching exercises.
Other: Relaxation — Diaphragmatic breathing will be taught as a relaxation exercise. The experimental group will be given both stretching and relaxation exercises. The Control group will be given only stretching exercises.
  Arms: The Experimental Group

SUMMARY:
The study aimed to examine the effect of stretching and relaxation exercises on pain and quality of life in women with primary dysmenorrhea.

DETAILED DESCRIPTION:
While dysmenorrhea is a frequent gynecologic condition that affects women of reproductive age, young women are generally unaware of it. Dysmenorrhea is divided into two main types based on its pathophysiology:

* Primary dysmenorrhea (PD), is menstrual discomfort coupled with regular ovulatory cycles and a defined physiological explanation. Adolescents and young adults are the most affected.
* Secondary dysmenorrhea (SD), is defined as menstruation discomfort caused by a disease (endometriosis, fibroids, adenomyosis, pelvic adhesions, endometrial polyps, pelvic inflammatory disease) or the use of an intrauterine contraceptive device.

Dysmenorrhea is a type of persistent, cyclic pelvic pain that can be accompanied by nausea, vomiting, diarrhea, headache, exhaustion, back pain, and dizziness. In studies conducted on university students in Turkey in 2009 and 2010, 87.7% and 72.7% (respectively) of the students reported that they had pain during the menstrual period.

The release of prostaglandins into the uterine tissue is assumed to be the cause of dysmenorrhea. As a result, nonsteroidal anti-inflammatory drugs (NSAIDs) are the usual first-line treatment for dysmenorrhea. Oral contraceptives, acupuncture, acupressure, yoga, and vitamin B1 are among the additional treatments that have been suggested.

It has been suggested that exercise can help with dysmenorrhea. Physical exercise has been suggested as a medical treatment for the treatment of dysmenorrhea and related symptoms by several writers. Billig was one of the first to advocate for exercise as a treatment for dysmenorrhea; he devised a set of stretching exercises and found a reduction in dysmenorrheic symptoms.

H1: There is a significant difference in pain and quality of life in the group with stretching and relaxation exercises compared to the group with stretching exercises.

ELIGIBILITY:
Inclusion Criteria:

* participants in the study voluntarily.
* participants in ages between 18-25 years of age.
* participants have a sedentary lifestyle.
* participant's pain intensity of more than 40 mm during the menstrual period according to the VAS.

Exclusion Criteria:

* using regular drugs like NSAIDs
* presence of SD
* having an irregular menstrual cycle
* presence of chronic disease.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 weeks
  Participants will be evaluated their menstrual pain levels on the Visual Analogue Scale between 0 and 10.
The Menstruation Symptom Questionnaire | 4 weeks
  Participants will rate their menstrual distress using the Menstrual Symptom Scale. The minimum score on this scale is 22, while the maximum score is 110. We can see that the lower the score in the questionnaire, the fewer problems the person has during the menstrual period.
Short Form 12 Health Survey | 4 weeks
  Participants will be evaluated their health-related quality of life using the Short Form 12 Health Survey. It is seen that the higher the score in the questionnaire, the higher the quality of life of the person.
Measurement with Algometer | 4 weeks
  Algometer measures the pain threshold, and in the study, it will be checked whether the pain thresholds changed with the exercises performed by the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Zöhre, Pt, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Ataşehir/İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferries-Rowe E, Corey E, Archer JS. Primary Dysmenorrhea: Diagnosis and Therapy. Obstet Gynecol. 2020 Nov;136(5):1047-1058. doi: 10.1097/AOG.0000000000004096. PMID 33030880
- [Background] Lopez-Liria R, Torres-Alamo L, Vega-Ramirez FA, Garcia-Luengo AV, Aguilar-Parra JM, Trigueros-Ramos R, Rocamora-Perez P. Efficacy of Physiotherapy Treatment in Primary Dysmenorrhea: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2021 Jul 23;18(15):7832. doi: 10.3390/ijerph18157832. PMID 34360122
- [Background] Proctor M, Farquhar C. Diagnosis and management of dysmenorrhoea. BMJ. 2006 May 13;332(7550):1134-8. doi: 10.1136/bmj.332.7550.1134. No abstract available. PMID 16690671
- [Background] Dorn LD, Negriff S, Huang B, Pabst S, Hillman J, Braverman P, Susman EJ. Menstrual symptoms in adolescent girls: association with smoking, depressive symptoms, and anxiety. J Adolesc Health. 2009 Mar;44(3):237-43. doi: 10.1016/j.jadohealth.2008.07.018. Epub 2008 Oct 29. PMID 19237109
- [Background] Petruzzello SJ, Landers DM, Hatfield BD, Kubitz KA, Salazar W. A meta-analysis on the anxiety-reducing effects of acute and chronic exercise. Outcomes and mechanisms. Sports Med. 1991 Mar;11(3):143-82. doi: 10.2165/00007256-199111030-00002. PMID 1828608
- [Background] Ameade EPK, Amalba A, Mohammed BS. Prevalence of dysmenorrhea among University students in Northern Ghana; its impact and management strategies. BMC Womens Health. 2018 Feb 13;18(1):39. doi: 10.1186/s12905-018-0532-1. PMID 29433488
- [Background] Bernardi M, Lazzeri L, Perelli F, Reis FM, Petraglia F. Dysmenorrhea and related disorders. F1000Res. 2017 Sep 5;6:1645. doi: 10.12688/f1000research.11682.1. eCollection 2017. PMID 28944048
- [Background] Kamel DM, Tantawy SA, Abdelsamea GA. Experience of dysmenorrhea among a group of physical therapy students from Cairo University: an exploratory study. J Pain Res. 2017 May 9;10:1079-1085. doi: 10.2147/JPR.S132544. eCollection 2017. PMID 28533696
- [Background] Burnett M, Lemyre M. No. 345-Primary Dysmenorrhea Consensus Guideline. J Obstet Gynaecol Can. 2017 Jul;39(7):585-595. doi: 10.1016/j.jogc.2016.12.023. PMID 28625286
- [Background] Doty E, Attaran M. Managing primary dysmenorrhea. J Pediatr Adolesc Gynecol. 2006 Oct;19(5):341-4. doi: 10.1016/j.jpag.2006.06.005. No abstract available. PMID 17060018
- [Background] Ryan SA. The Treatment of Dysmenorrhea. Pediatr Clin North Am. 2017 Apr;64(2):331-342. doi: 10.1016/j.pcl.2016.11.004. PMID 28292449
- [Background] Granot M, Yarnitsky D, Itskovitz-Eldor J, Granovsky Y, Peer E, Zimmer EZ. Pain perception in women with dysmenorrhea. Obstet Gynecol. 2001 Sep;98(3):407-11. doi: 10.1016/s0029-7844(01)01465-x. PMID 11530120
- [Background] Tu CH, Niddam DM, Chao HT, Chen LF, Chen YS, Wu YT, Yeh TC, Lirng JF, Hsieh JC. Brain morphological changes associated with cyclic menstrual pain. Pain. 2010 Sep;150(3):462-468. doi: 10.1016/j.pain.2010.05.026. PMID 20705214
- [Background] French L. Dysmenorrhea in adolescents: diagnosis and treatment. Paediatr Drugs. 2008;10(1):1-7. doi: 10.2165/00148581-200810010-00001. PMID 18162003
- [Background] Yu A. Complementary and alternative treatments for primary dysmenorrhea in adolescents. Nurse Pract. 2014 Nov 16;39(11):1-12. doi: 10.1097/01.NPR.0000454984.19413.28. PMID 25325520
- [Background] Xu K, Chen L, Fu L, Xu S, Fan H, Gao Q, Xu Y, Wang W. Stressful Parental-Bonding Exaggerates the Functional and Emotional Disturbances of Primary Dysmenorrhea. Int J Behav Med. 2016 Aug;23(4):458-63. doi: 10.1007/s12529-015-9504-0. PMID 26309099
- [Background] ACOG Committee Opinion No. 760: Dysmenorrhea and Endometriosis in the Adolescent. Obstet Gynecol. 2018 Dec;132(6):e249-e258. doi: 10.1097/AOG.0000000000002978. PMID 30461694
- [Background] Morrow C, Naumburg EH. Dysmenorrhea. Prim Care. 2009 Mar;36(1):19-32, vii. doi: 10.1016/j.pop.2008.10.004. PMID 19231600
- [Background] Marjoribanks J, Ayeleke RO, Farquhar C, Proctor M. Nonsteroidal anti-inflammatory drugs for dysmenorrhoea. Cochrane Database Syst Rev. 2015 Jul 30;2015(7):CD001751. doi: 10.1002/14651858.CD001751.pub3. PMID 26224322
- [Background] Pattanittum P, Kunyanone N, Brown J, Sangkomkamhang US, Barnes J, Seyfoddin V, Marjoribanks J. Dietary supplements for dysmenorrhoea. Cochrane Database Syst Rev. 2016 Mar 22;3(3):CD002124. doi: 10.1002/14651858.CD002124.pub2. PMID 27000311
- See also: Health definition according to World Health Organization — https://www.who.int/data/gho/data/major-themes/health-and-well-being